CLINICAL TRIAL: NCT06152198
Title: Internal Fixation Versus Hip Replacement in Older Adults with an Garden I/II Femoral Neck Fracture: Physical Function and Pain in Elderly Patients - a Substudy of the Hipsther Trial
Brief Title: Functional Outcome After ORIF or Arthroplasty for Femoral Neck Fracture
Acronym: HipFunct
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hipsther hip function
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Hip Fractures; Femoral Neck Fractures; Undisplaced Fracture; Treatment Complication; Internal Fixation; Complications; Arthroplasty Complications
Keywords: hip fracture; femoral neck fracture; treatment; hip arthroplasty; internal fixation
MeSH Terms: conditions — Hip Fractures; Femoral Neck Fractures | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hip arthroplasty (Experimental): Operative treatment with hip arthroplasty i.e cemented total- or hemiarthroplasty.
  Interventions: Device: Treatment
- Internal fixation (Active Comparator): Operative treatment with internal fixation i.e screws, pins, hook pins, sliding hip device.
  Interventions: Device: Treatment

INTERVENTIONS:
Device: Treatment — Allocation to hip arthroplasty or internal fixation. The choice between hemi- or total hip arthroplasty in the arthroplasty group and type of osteosynthesis are the surgeon preference.

SUMMARY:
Aim To investigate the effect of internal fixation versus hip arthroplasty on physical function and pain in elderly patients.

Methods This is a substudy of an on-going nationwide multicenter registry-based RCT named HipSTHeR- (Hip Screws or Total Hip replacement or undisplaced femoral neck fracture in elderly patients) [21]. The aim is to recruit 340 patients with undisplaced or minimally displaced femoral neck fracture, Garden 1 or 2, are randomized to surgery either with internal screw fixation or hip arthroplasty.

This substudy aims to investigate the potential differences between internal fixation versus hip arthroplasty regarding physical function and pain 4- and 12- months after surgery. Those included in the main study will be contacted by letter a few weeks after the surgery to be invited to participate in a further study. The assessor will then contact the person by telephone to answer further questions and to obtain informed consent. The follow-ups will be conducted over telephone and mail at 4 and 12 months. During the follow-up the participants will answer questions about their functional level.

Information on randomisation and fracture data will be acquired from the Swedish Fracture Register and treatment data from the Swedish Hip Arthroplasty Register.

Primary outcome The New Mobility Score will be used as the primary outcome with follow-up at 4- and 12 months.

Secondary outcome WOMAC will be used as an additional hip specific patient reported outcome.

Activities of daily living will be assessed with Katz ADL index to evaluate the patients' performance and the need of assistance in ADL.

Patients' cognitive status will be assessed ALFI-MMSE, adapted from Adult Lifestyles and Function Interview (ALFI-MMSE).

The Geriatric Depression Scale (GDS-15), which are developed to identify depressive symptoms.

The Philadelphia Geriatric Center Morale Scale (PGCMS) and have been used in several studies including frail people living in residential care facilities and can be used among patients with cognitive impairment.

DETAILED DESCRIPTION:
Aim To investigate the effect of internal fixation versus hip arthroplasty on physical function and pain in elderly patients.

Methods This is a substudy of an on-going nationwide multicenter registry-based RCT named HipSTHeR- (Hip Screws or Total Hip replacement or undisplaced femoral neck fracture in elderly patients) [21]. Patients with undisplaced or minimally displaced femoral neck fracture, Garden 1 or 2, are randomized to surgery either with internal screw fixation or hip arthroplasty.

This substudy aims to investigate the potential differences between internal fixation versus hip arthroplasty regarding physical function and pain 4- and 12- months after surgery. Those included in the main study will be contacted by letter a few weeks after the surgery to be invited to participate in a further study. The assessor will then contact the person by telephone to answer further questions and to obtain informed consent. The follow-ups will be conducted over telephone and mail at 4 and 12 months. During the follow-up the participants will answer questions about their functional level.

The inclusion criteria for the Hipsther trial are: >75 years and an undisplaced or minimally displaced femoral neck fracture, classified as Garden I or II on conventional radiograph, eligible for internal fixation and hip arthroplasty and treatment at participating unit. The exclusion criteria are pathological or stress fractures, peri-implant femoral neck fracture and previous inclusion of a contralateral Garden 1 or 2 femoral neck fracture. Patients with cognitive impairment are also included. The inclusion criteria for this substudy is inclusion in the Hipsther trial and the participants require a functional language in Swedish.

Information on randomisation and fracture data will be acquired from the Swedish Fracture Register and treatment data from the Swedish Hip Arthroplasty Register.

Primary outcome The New Mobility Score will be used as the primary outcome with follow-up at 4- and 12 months. The New Mobility Score is an evaluation of patient's ability to perform: walking indoor, outdoor and shopping. Each item is scored between 0 and 3 (0: not at all, 1: with help from another person, 2: with an aid, 3: no difficulty) resulting in a total of 9 points. The New Mobility Score (NMS) may predict mortality, predict function and has a high inter-tester reliability.

Secondary outcome WOMAC will be used as an additional hip specific patient reported outcome. The scale contains 24 items; divided in pain, stiffness and physical function, on a scale of 0 to 4, where lower score indicates a lower level of symptom and physical disability. WOMAC has been found to have good reliability and validity in elderly patients with femoral neck fracture and is widely used in the evaluation of hip osteoarthritis. The patients' pain will also be assessed with NRS, both in rest and activity. WOMAC will be assessed at 4- and 12 months follow-up.

Activities of daily living will be assessed with Katz ADL index to evaluate the patients' performance and the need of assistance in ADL. The Katz ADL index measures both Personal-ADL (P-ADL, bathing, dressing, toileting, transfer, continence and feeding) and Instrumental ADL (I-ADL, cleaning, shopping, transportation, and cooking), higher scores indicating greater ADL dependence.

Patients' cognitive status will be assessed ALFI-MMSE, adapted from Adult Lifestyles and Function Interview (ALFI-MMSE). To discover depressive symptoms, we will use The Geriatric Depression Scale (GDS-15), which are developed to identify depressive symptoms with 15 "yes" or "no" questions, and higher scores indicating greater depressive symptoms. The participants subjective well-being or morale will be assessed with The Philadelphia Geriatric Center Morale Scale (PGCMS) and have been used in several studies including frail people living in residential care facilities and can be used among patients with cognitive impairment. The PGCMS has 17 dichotomized items, and the scores vary between 0 to 17, where a high morale is described as a basic sense of satisfaction with oneself and according to the instructions scores 0-9 indicates a low morale, 10-12 indicates intermediate and 13-17 high morale.

Sample size The sample size calculation was performed similarly to the Sense trial [34]. We assumed a minimal clinically important difference in NMS of 1 point and a 1-year average of 6.4 points with an SD of 2.2 [35]. Assuming a 1-point difference with an SD of 2.2, allowing a 5% probability of type 1 error for a 95% statistical power. 127 patients are required in each group. To allow for loss during follow-up due to mortality and internal dropout (25%). Therefore, a total of 340 patients are required for the study.

ELIGIBILITY:
Inclusion Criteria:

* Undisplaced (Garden I-II) femoral neck fracture (within 72h)
* Treated at participating unit
* Informed consent
* Amenable for both treatment options
* Included in the Hipsther trial

Exclusion Criteria:

* No informed consent
* Pathological or stress fracture
* Peri-implant fracture
* Previous inclusion of a contralateral Garden 1 or 2 femoral neck fracture

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2021-06-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
New Mobility Score | 4- and 12 months
  The New Mobility Score is an evaluation of patient's ability to perform: walking indoor, outdoor and shopping. Each item is scored between 0 and 3 (0: not at all, 1: with help from another person, 2: with an aid, 3: no difficulty) resulting in a total of 9 points.

SECONDARY OUTCOMES:
WOMAC | 4- and 12 months
  An additional hip specific patient reported outcome. The scale contains 24 items; divided in pain, stiffness and physical function, on a scale of 0 to 4, where lower score indicates a lower level of symptom and physical disability [25]. WOMAC has been found to have good reliability and validity in elderly patients with femoral neck fracture [26] and is widely used in the evaluation of hip osteoarthritis. The patients' pain will also be assessed with NRS, both in rest and activity.
Katz ADL index | 4- and 12 months
  Activities of daily living will be assessed with Katz ADL index to evaluate the patients' performance and the need of assistance in ADL. The Katz ADL index measures both Personal-ADL (P-ADL, bathing, dressing, toileting, transfer, continence and feeding) and Instrumental ADL (I-ADL, cleaning, shopping, transportation, and cooking), higher scores indicating greater ADL dependence.
ALFI-MMSE | 4- and 12 months
  Patients' cognitive status will be assessed ALFI-MMSE, adapted from Adult Lifestyles and Function Interview (ALFI-MMSE) [28]. To discover depressive symptoms, we will use The Geriatric Depression Scale (GDS-15) [29], which are developed to identify depressive symptoms with 15 "yes" or "no" questions, and higher scores indicating greater depressive symptoms.
Philadelphia Geriatric Center Morale Scale (PGCMS) | 4- and 12 months
  The participants subjective well-being or morale will be assessed with The Philadelphia Geriatric Center Morale Scale (PGCMS) and have been used in several studies including frail people living in residential care facilities and can be used among patients with cognitive impairment. The PGCMS has 17 dichotomized items, and the scores vary between 0 to 17, where a high morale is described as a basic sense of satisfaction with oneself and according to the instructions scores 0-9 indicates a low morale, 10-12 indicates intermediate and 13-17 high morale.

CONTACTS AND LOCATIONS:
Overall Officials: Olof Wolf, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Olof Wolf, Uppsala, Sweden

REFERENCES:
- [Background] Wolf O, Sjoholm P, Hailer NP, Moller M, Mukka S. Study protocol: HipSTHeR - a register-based randomised controlled trial - hip screws or (total) hip replacement for undisplaced femoral neck fractures in older patients. BMC Geriatr. 2020 Jan 21;20(1):19. doi: 10.1186/s12877-020-1418-2. PMID 31964340
- [Background] Mukka S, Sjoholm P, Aziz A, Eisler T, Kadum B, Krupic F, Morberg P, Sayed-Noor A. A cohort study comparing internal fixation for undisplaced versus hip arthroplasty for displaced femoral neck fracture in the elderly: a pilot study for a clinical trial. Pilot Feasibility Stud. 2020 Jul 11;6:98. doi: 10.1186/s40814-020-00642-w. eCollection 2020. PMID 32670600
- [Background] Parker MJ, Palmer CR. A new mobility score for predicting mortality after hip fracture. J Bone Joint Surg Br. 1993 Sep;75(5):797-8. doi: 10.1302/0301-620X.75B5.8376443.
- [Background] Burgers PT, Poolman RW, Van Bakel TM, Tuinebreijer WE, Zielinski SM, Bhandari M, Patka P, Van Lieshout EM; HEALTH and FAITH Trial Investigators. Reliability, validity, and responsiveness of the Western Ontario and McMaster Universities Osteoarthritis Index for elderly patients with a femoral neck fracture. J Bone Joint Surg Am. 2015 May 6;97(9):751-7. doi: 10.2106/JBJS.N.00542. PMID 25948522
- [Background] Viberg B, Kold S, Brink O, Larsen MS, Hare KB, Palm H; SENSE collaborators. Is arthroplaSty bEtter than interNal fixation for undiSplaced femoral nEck fracture? A national pragmatic RCT: the SENSE trial. BMJ Open. 2020 Oct 10;10(10):e038442. doi: 10.1136/bmjopen-2020-038442. PMID 33040011